CLINICAL TRIAL: NCT06905132
Title: Preoperative 5-Day Radiotherapy for Soft Tissue Sarcoma: A Single Institution Phase II Trial
Brief Title: Preoperative 5-Day Radiotherapy for Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jennifer Lynn Harper, Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104131; Pro00141818 (Other: Medical University of South Carolina)
Record Dates: First submitted 2025-03-12; First posted 2025-04-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: STS; HFRT; SFRP2
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypofractionated Radiation Therapy (Experimental)
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Participants will receive preoperative 5-day HFRT (30Gy/5fx once daily over consecutive weekdays) followed by "standard of care" wide local excision 2-6 weeks later.

SUMMARY:
The purpose of this research study is to preserve healthy tissue around the cancer on the arm(s) and/or leg(s) using Hypofractionated radiotherapy, while treating the cancer and preventing it from spreading to other areas of the body.

DETAILED DESCRIPTION:
This study is for subjects that have been diagnosed with cancer in their arm, leg, or trunk (the part of the body that involves the chest, abdomen, and pelvis). The purpose of this research study is to preserve healthy tissue around the cancer on the arm(s) and/or leg(s) using Hypofractionated radiotherapy, while treating the cancer and preventing it from spreading to other areas of the body. This study will look at early side effects and effectiveness of preoperative 5-day Hypofractionated radiotherapy. Active participation in the study will take about 12 visits and are completed once the participant has a 6-month post-operation visit.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and provision of informed consent via signed and dated copy.
* Histologically confirmed STS of extremity or trunk.
* Male or female, aged greater than or equal to 18 years old
* ECOG performance status 0-3
* Meets screening criteria for receipt of radiotherapy.
* Deemed eligible for wide local excision.
* Patient and/or physician identified possible barriers to receiving a 5-week course of conventionally fractionated preoperative radiotherapy. Potential barriers include but are not limited to concern for local progression that could precluded or complicate limb sparing surgery, concern for distant progression that could result in patient being non-operative, financial and/or physical burden of travel for daily treatments, financial burden of time away from work or caregiving.

Exclusion Criteria:

* Distant metastatic disease
* Prior radiation therapy in the proposed treatment area
* Simultaneous treatment of another malignancy
* Women who are pregnant or plan to become pregnant during the period of radiation therapy
* Planned concurrent administration of chemotherapy and radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
HFRT Safety | 6 months
  Evaluate the safety of 5-day HFRT as measured by the rates of major wound complications occurring within 120 days of surgery.

SECONDARY OUTCOMES:
Treatment Response | 6 months
  Evaluate treatment response to 5-day HFRT as measured by pathologic response. Pathologic response is defined as percent necrosis and percent viable tumor.
Safety Profile | 6 months
  Evaluate the safety profile of 5-day HFRT, specifically the proportion of patients experiencing acute toxicities and late toxicities

OTHER OUTCOMES:
Control Rate | 3 years
  Estimate 3-year local control rate of 5-day HFRT
Relapse-free Survival | 3 years
  Estimate 3-year relapse-free survival. Relapse-free survival is defined as the time from surgery to disease recurrence or death from any cause. 3-year overall survival of 5-day HFRT
Overall Survival | 3 years
  3-year overall survival of 5-day HFRT. Overall survival is defined as the time from RT initiation to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Harper, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States